CLINICAL TRIAL: NCT03156062
Title: Climatotherapy at Red Sea - Hurghada Versus Topical Combination of Corticosteroids and Salicylic Acid in Treatment of Psoriasis
Brief Title: Climatotherapy Versus Topical Combination of Corticosteroids and Salicylic Acid in Treatment of Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ESAhmed, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CCS
Record Dates: First submitted 2017-05-13; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Papulosquamous Skin Disease
MeSH Terms: conditions — Skin Diseases, Papulosquamous | interventions — Adrenal Cortex Hormones; Salicylic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Drug: Topical corticosteroids with salicylic acid
- control group (Active Comparator)
  Interventions: Drug: Topical corticosteroids with salicylic acid

INTERVENTIONS:
Drug: Topical corticosteroids with salicylic acid — comparison between climatotherapy and topical combination of corticosteroids and salicylic acid in treatment of psoriasis

SUMMARY:
Psoriasis is a multisystem disease predominately manifested as chronic inflammation of the skin and characterized by scaly, erythematous patches, papules and plaques, which are often pruritic. As chronic disease, psoriasis waxes and wanes throughout patient life time. The disease course is modified with initiation and cessation of treatment, and spontaneous remission is rare. Clinically lesions can be distributed in any part of the body, this leads to impaired consequences on the perception of body image, social relations and in general on quality of life.

DETAILED DESCRIPTION:
The severity of psoriasis is defined by the extent of body surface involvement as well as the involvement of areas that substantially affect daily life such as hands, feet, face and genital region . Approximately 80% of patients have mild to moderate disease and 20% have moderate to severe disease. Although the precise etiology of psoriasis remains unknown, a combination of immunologic, genetic and environmental factors contribute to its development and exacerbation. Psoriasis has multifactorial pathogenesis in which predisposing genetic factors (dysregulation of the immune system and alteration of keratinocytes) and environmental trigger factors (such as local trauma, streptococcal infections, emotional stress, drugs as B-blockers and lithium) interact with each other by triggering a specific immune response mediated by T-lymphocytes.Treatment of psoriasis is still very complex. Several treatments for plaque psoriasis are available as topical medications for mild to moderate cases of psoriasis (corticosteroids, vit D3 analogues, salicylic acid, dithranol etc.). Phototherapy is useful in moderately-severe psoriasis unresponsive to topical therapy alone. Systemic treatment is used for severe forms of psoriasis including immunosuppressive drugs such as methotrexate or cyclosporine, retinoids, etc., and in cases of contraindications or ineffectiveness of these drugs these severe forms of psoriasis can be treated with biological drugs such as adalimumab, etanercept, infliximab, etc.The climatotherapy presents a safe and efficient alternative to conventional therapeutic modality for psoriasis. Climatotherapy treatment is based on healing capacities of natural resources.Climatic treatment includes balneotherapy and sun exposure. Balneotherapy represents a set of methods and practices (bathing, drinking, inhalation, etc.)

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of psoriasis(mild to moderate) .
2. Age 9-60 years

Exclusion Criteria:

1-Patients under 9 years. 2-Patient with severe psoriasis. 3-Skin cancer. 4-Renal insufficiency. 5-Acute infections. 6-Severe hypertension. 7-Skin and systemic diseases worsened by sun exposure. 8-Acute and non controlled concomitant diseases. 9-Ischemic heart diseases or any disease rendering them unable to bathe.

Ages: 9 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-10-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Good response to treatment | 1day
  Didital photography and histopathalogical examination

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naldi L, Gambini D. The clinical spectrum of psoriasis. Clin Dermatol. 2007 Nov-Dec;25(6):510-8. doi: 10.1016/j.clindermatol.2007.08.003. PMID 18021886
- [Background] American Academy of Dermatology Work Group; Menter A, Korman NJ, Elmets CA, Feldman SR, Gelfand JM, Gordon KB, Gottlieb A, Koo JY, Lebwohl M, Leonardi CL, Lim HW, Van Voorhees AS, Beutner KR, Ryan C, Bhushan R. Guidelines of care for the management of psoriasis and psoriatic arthritis: section 6. Guidelines of care for the treatment of psoriasis and psoriatic arthritis: case-based presentations and evidence-based conclusions. J Am Acad Dermatol. 2011 Jul;65(1):137-74. doi: 10.1016/j.jaad.2010.11.055. Epub 2011 Feb 8. PMID 21306785
- [Background] Bowcock AM, Cookson WO. The genetics of psoriasis, psoriatic arthritis and atopic dermatitis. Hum Mol Genet. 2004 Apr 1;13 Spec No 1:R43-55. doi: 10.1093/hmg/ddh094. PMID 14996755
- [Background] Harari M, Czarnowicki T, Fluss R, Ruzicka T, Ingber A. Patients with early-onset psoriasis achieve better results following Dead Sea climatotherapy. J Eur Acad Dermatol Venereol. 2012 May;26(5):554-9. doi: 10.1111/j.1468-3083.2011.04099.x. Epub 2011 May 17. PMID 21575063
- [Background] Harari M, Novack L, Barth J, David M, Friger M, Moses SW. The percentage of patients achieving PASI 75 after 1 month and remission time after climatotherapy at the Dead Sea. Int J Dermatol. 2007 Oct;46(10):1087-91. doi: 10.1111/j.1365-4632.2007.03278.x. PMID 17910722
- [Background] Chren MM, Lasek RJ, Quinn LM, Mostow EN, Zyzanski SJ. Skindex, a quality-of-life measure for patients with skin disease: reliability, validity, and responsiveness. J Invest Dermatol. 1996 Nov;107(5):707-13. doi: 10.1111/1523-1747.ep12365600. PMID 8875954
- [Background] Fredriksson T, Pettersson U. Severe psoriasis--oral therapy with a new retinoid. Dermatologica. 1978;157(4):238-44. doi: 10.1159/000250839. PMID 357213
- [Background] Guenther LC. Fixed-dose combination therapy for psoriasis. Am J Clin Dermatol. 2004;5(2):71-7. doi: 10.2165/00128071-200405020-00001. PMID 15109271
- [Background] Gottlieb A, Korman NJ, Gordon KB, Feldman SR, Lebwohl M, Koo JY, Van Voorhees AS, Elmets CA, Leonardi CL, Beutner KR, Bhushan R, Menter A. Guidelines of care for the management of psoriasis and psoriatic arthritis: Section 2. Psoriatic arthritis: overview and guidelines of care for treatment with an emphasis on the biologics. J Am Acad Dermatol. 2008 May;58(5):851-64. doi: 10.1016/j.jaad.2008.02.040. PMID 18423261